CLINICAL TRIAL: NCT01426178
Title: Neurally Adjusted Ventilatory Assist (NAVA) in NonInvasive Ventilation (NIV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0099
Record Dates: First submitted 2011-07-07; First posted 2011-08-31 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory Insufficiency; Respiration, Artificial; Intermittent Positive-Pressure Ventilation; Neurally Adjusted Ventilatory Assist; Non Invasive Ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration | interventions — Interactive Ventilatory Support; Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist in Non Invasive Ventilation (Device) — After written information and consent, patients are randomised in two groups: NAVA first or PSV first.
  They receive a NAVA catheter, which has exactly the same appearance as a standard naso-gastric catheter.

SUMMARY:
Main hypothesis is that Neurally Adjusted Ventilatory Assist (NAVA) allows asynchrony reduction in non invasive ventilation (NIV) in comparison with reference Pressure Support (PSV) mode.

The purpose of the protocol is to compare asynchrony rate between periods of pressure support and periods of NAVA.

DETAILED DESCRIPTION:
After written information and consent, patients are randomised in two groups: NAVA first or PSV first.

They receive a NAVA catheter, which has exactly the same appearance as a standard naso-gastric catheter.

A standardised set of 1 hour of non-invasive ventilation is started. Depending on the randomisation group, patients start with a 30 minutes set of NIV with NAVA settings or with a 30 minutes set of NIV with PSV settings. A 30-minute watch-out period is then delivered with no mechanical ventilation.

Then a second 30-minute set of NIV in the other settings (NAVA or PSV depending on the randomisation) is delivered.

During each set of NIV, flow, volume, pressure and EADi are recorded during 10 minutes, after a 10-minute period of equilibration. Recordings will be processed by two blind investigators in order to count the number of asynchronies. In case of disagreement between investigators, a third one will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* - Patient older then 18 years
* Patient requiring first non invasive ventilation set because of acute respiratory failure

Exclusion Criteria:

* Patients protected by the law
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Asynchrony rate defined as a percentage of the total respiratory rate | at 90 minutes

SECONDARY OUTCOMES:
- Number of patients presenting a high asynchrony rate (>10%) | at 90 minutes
Oxygenation evaluated as the PaO2 / FiO2 ratio at the end of considered NAVA set | at 90 minutes
Patient comfort | at 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bertrand PM, Futier E, Coisel Y, Matecki S, Jaber S, Constantin JM. Neurally adjusted ventilatory assist vs pressure support ventilation for noninvasive ventilation during acute respiratory failure: a crossover physiologic study. Chest. 2013 Jan;143(1):30-36. doi: 10.1378/chest.12-0424. PMID 22661448